CLINICAL TRIAL: NCT04263480
Title: Efficacy and Safety of Carfilzomib in Combination With Ibrutinib vs Ibrutinib Alone in Waldenström's Macroglobulinemia (CZAR-1)
Brief Title: Efficacy and Safety of Carfilzomib in Combination With Ibrutinib vs Ibrutinib in Waldenström's Macroglobulinemia
Acronym: CZAR-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christian Buske (Other)
Collaborators: Amgen (Industry); Janssen, LP (Industry)
Responsible Party: Sponsor-Investigator, Christian Buske, Prof. Dr. med., University of Ulm
Organization: University of Ulm (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZAR-1
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: MYD88 mutation; CXCR4 mutation; Carfilzomib; Ibrutinib; Hematology; Oncology
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Neoplasms | interventions — carfilzomib; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Carfilzomib + Ibrutinib (Experimental): Patients will be treated with Ibrutinib until evidence of progressive disease or no longer tolerated. Patients will receive in addition Carfilzomib for two years.
  Interventions: Drug: Carfilzomib + Ibrutinib
- Arm B: Ibrutinib (Active Comparator): Patients will be treated with Ibrutinib until evidence of progressive disease or no longer tolerated.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Carfilzomib + Ibrutinib — Carfilzomib:
  Cycle 1, day 1: 20 mg/m² i.v. Cycle 1, day 8, day 15: 70 mg/m² i.v. Cycle 2 - 12, day 1, day 8, day 15: 70 mg/m² i.v. Cycle 13 - 24, day 1, day 15: 70 mg/m² i.v.
  Ibrutinib:
  420 mg p.o daily until disease progression or non-tolerable toxicities
  Arms: Arm A: Carfilzomib + Ibrutinib
Drug: Ibrutinib — Ibrutinib:
  420 mg p.o daily until disease progression or non-tolerable toxicities
  Arms: Arm B: Ibrutinib

SUMMARY:
In Waldenström macroglobulinemia (WM) chemotherapy induces only low CR/VGPR (Complete Remission/ Very Good Partial Response) rates and responses of short duration compared to other indolent lymphomas. Thus, innovative approaches are needed which combine excellent activity and tolerability in WM. Chemotherapy-free approaches are highly attractive for this patient group. Based on its high activity in WM and its low toxicity, Ibrutinib was approved for the treatment of WM by the European Medicines Agency (EMA). However, also Ibrutinib fails to induce CRs and the VGPR rate is 16% in relapsed patients. In addition, activity of Ibrutinib depends on the genotype: compared to MYD88mut/CXCR4WT patients Ibrutinib single agent therapy induces substantially lower response rates in patients with the MYD88mut/CXCR4mut or the MYD88WT/CXCR4WT genotype (major response (at least PR) in 91.7 % compared to 61.9 and 0 %, respectively). Phase II data have indicated that the proteasome inhibitor Carfilzomib is able to overcome the inferior prognosis of Ibrutinib in MYD88mut/CXCR4mut and MYD88WT/CXCR4WT patients, as response rates were high for all genotypes in a phase II study combining Carfilzomib with Rituximab and Dexamethasone. Based on this the investigators hypothesize that addition of Carfilzomib to Ibrutinib will increase the VGPR/CR rate compared to Ibrutinib alone in patients with WM, in particular in patients carrying the CXCR4 mutation. In addition, the investigators hypothesize, that the combination Carfilzomib and Ibrutinib will be also highly active in MYD88 wildtype patients and that this combination will be at least as efficient in treatment naïve patients as in relapsed/refractory patients.

DETAILED DESCRIPTION:
In Waldenström macroglobulinemia (WM) conventional chemotherapy induces only low Complete Remission (CR) rates and responses of short duration compared to other indolent lymphomas. Thus, innovative approaches are needed which combine excellent activity and tolerability in patients with WM, who are mostly of advanced age. Today, chemotherapy in combination with the anti-CD20 antibody Rituximab is still the backbone of treatment in patients with WM and is recommended as first line in national and international treatment guidelines.With the approval of Ibrutinib by the EMA 2015 for patients with relapsed WM or for patients not eligible for chemotherapy with treatment naïve WM treatment landscape has changed in this lymphoma subtype and there is an urgent need to evaluate to which extent chemotherapy-free approaches add clinical benefit to the patient. Based on its high activity in WM and its low toxicity, Ibrutinib was approved for the treatment of WM by the EMA. However, also Ibrutinib fails to induce CRs and the VGPR (Very Good Partial Response) rate is 16% in relapsed patients. In addition, activity of Ibrutinib depends on the genotype with inferior response rates in MYD88mut/CXCR4mut patients and in patients with unmutated MYD88 and CXCR4 compared to MYD88mut/CXCR4WT patients (major response (at least PR) in 91.7 % compared to 61.9 and 0 %, respectively). Phase II data have indicated that the proteasome inhibitor Carfilzomib is able to overcome the inferior prognosis of Ibrutinib in MYD88mut/CXCR4mut and MYD88WT/CXCR4WT patients, as response rates were high for all genotypes in a phase II study combining Carfilzomib with Rituximab and Dexamethasone. Based on this the investigators hypothesize that addition of Carfilzomib to Ibrutinib will increase the VGPR/CR rate compared to Ibrutinib alone in patients with WM, in particular in patients carrying the CXCR4 mutation. In addition, the investigators hypothesize, that the combination Carfilzomib and Ibrutinib will be also highly active in MYD88 wildtype patients and that this combination will be at least as efficient in treatment naïve patients as in relapsed/refractory patients.

The study is an international, phase II, multicenter, open label and randomized trial comparing Carfilzomib in combination with Ibrutinib (treatment Arm A) versus Ibrutinib (treatment arm B) in male or female patients aged ≥ 18 years of de novo and relapsed/refractory WM in need of treatment.

The phase II study will consist of an open labeled, stratified 1:1 randomization between Arm A and Arm B. Stratification factors are MYD88 and CXCR4 status (positive vs. negative) and number of prior lines (0 vs. ≥ 1 treatment lines). A stratified central block randomization will be used.

The primary objective of the trial is to test the efficacy and toxicity of Carfilzomib and Ibrutinib in patients with treatment naïve or relapsed WM.

The aim of this study is to investigate the rate of CR or VGPR 12 months after the start of treatment using the response criteria updated at the Sixth IWWM (CR/VGPR).

99 patients at approximately 25 investigator sites will be recruited. Patients will be followed up after end of treatment. Patients will receive Ibrutinib in both treatment arms until progression, non-tolerated toxicity or until the study duration has reached its maximum of 7 years after the first patient was included into the trial. Follow-up (5 years or until disease progression for patients who discontinue treatment due to toxicity) or survival follow-up (for patients with progression disease) will be performed until the study duration has reached its maximum of 7 years after the first patient was included into the trial.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in this study:

* Proven clinicopathological diagnosis of WM as defined by consensus panel one of the Second International Workshop on WM. Histopathology has to occur before randomization within the last 4 months. In addition, pathological specimens have to be sent to the pathological reference center prior to randomization for the determination of the mutational status of MYD88 and CYCR4. Immunophenotyping will be performed in each center and saved locally. The positivity for CD20 can be assumed from any previous bone marrow immunohistochemistry or flow cytometry analysis performed up to 4 months prior to enrollment. Flow cytometry of bone marrow and blood cells will include at least one double staining and assess the disease specific expressions.
* De novo and relapsed/refractory WM independent of the genotype.
* Determination of mutational status of MYD88 and CXCR4.
* Patients must have at least one of the following criteria to initiate treatment as partly defined by "Consensus Panel Two" recommendations from the Second International Workshop on Waldenström Macroglobulinemia:

  * Recurrent fever, night sweats, weight loss, fatigue (at least one of them).
  * Hyperviscosity.
  * Lympadenopathy which is either symptomatic or bulky (≥ 5 cm in maximum diameter).
  * Symptomatic hepatomegaly and/or splenomegaly.
  * Symptomatic organomegaly and/or organ or tissue infiltration.
  * Peripheral neuropathy due to WM.
  * Symptomatic cryoglobulinemia.
  * Cold agglutinin anemia.
  * IgM related immune hemolytic anemia and/or thrombocytopenia.
  * Nephropathy related to WM.
  * Amyloidosis related to WM.
  * Hemoglobin ≤ 10 g/dL (patients should not have received red blood cells transfusions for at least 7 days prior to obtaining the screening haemoglobin).
  * Platelet count < 100 x 109/L (caused by BM infiltration of the lymphoma).
  * Serum monoclonal protein > 5 g/dL, even with no overt clinical symptoms.
  * IgM serum concentration ≥ 5g/dl.
  * and other WM associated relevant symptoms.
* World Health Organization (WHO)/ECOG performance status 0 to 2.
* Left ventricular ejection fraction ≥ 40% as assessed by transthoracic echocardiogram (TTE).
* Other criteria

  * Age ≥ than 18 years (male and female).
  * Life expectancy > 3 months.
  * Baseline platelet count ≥ 50 x 109/L, absolute neutrophil count ≥ 0.75 x 109/L. (if not due to BM infiltration by the lymphoma).
  * Meet the following pre-treatment laboratory criteria at the Screening visit conducted within 30 days prior to randomization:
* ASAT (SGPOT): < 3.0 times the ULN.
* ALAT (SGPT): < 3.0 times the ULN.
* Total Bilirubin: < 1.5 times the ULN, unless clearly related to the disease (except if due to Gilbert's syndrome).
* Serum creatinine: ≤ 2 mg/dl.
* Women of childbearing potential (WOCBP) must agree to use a highly effective method of birth control for the duration of the therapy up to 6 months after end of therapy. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner or sexual abstinence. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. Contraception and pregnancy testing are required according the CTFG recommendations.
* Men must agree not to father a child for the duration of therapy and 6 months after (use of a condom) and must agree to advice a female partner to use a highly effective method of birth control. Males must refrain from sperm donation for at least 6 months after the last dose of treatment.
* Voluntary written informed consent in the native language of the patient before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrolment:

* Previous treatments with following substances:

  * Prior exposure to Ibrutinib or other BTK inhibitors.
  * Prior exposure to Carfilzomib. Prior exposure to other proteasome inhibitors is allowed if the patients were not refractory, that is, had a remission (at least minor response) duration of ≥ 6 months. Prior plasmapheresis and short-term administration of corticosteroids ≤ 6 weeks administered at a dose equivalent to ≤ 20 mg/day of prednisone is also allowed.
* Serious medical or psychiatric illness (especially undergoing treatment) likely to interfere with participation in this clinical study.
* Active HIV, HBV or HCV infection.
* Central Nervous System involvement by lymphoma.
* History of a non-lymphoid malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate specific antigen for ≥ 1 year prior to randomization, other Stage 1 or 2 cancer treated with a curative intent and currently in complete remission, for ≥ 3 years.
* Uncontrolled illness including, but not limited to:

  * Uncontrolled diabetes mellitus (as indicated by metabolic derangements and / or severe diabetes mellitus related uncontrolled organ complications).
  * Chronic symptomatic congestive heart failure (Class NYHA III or IV) or LVEF < 40%.
  * Unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months prior to randomization.
  * Clinically significant cardiac arrhythmia that is symptomatic or requires treatment, or asymptomatic sustained ventricular tachycardia.
  * Known pericardial disease.
  * Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
  * Cardiac amyloidosis.
* Recent major surgery within 30 days prior to randomization.
* Known cirrhosis (meeting child-pugh stage C).
* Approved or investigational anticancer treatment within 21 days prior to randomization.
* Glucocorticoid therapy within 14 days prior to randomization that exceeds a cumulative dose of 160 mg of Dexamethasone or equivalent dose of other corticosteroids.
* Focal radiation therapy within 7 days prior to randomization. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to randomization (i.e. prior radiation must have been to less than 30% of the bone marrow).
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs.
* Hypersensitivity to the active substances or to any of the excipients of the investigational medicinal products.
* Active infection within 14 days prior to randomization requiring systemic antibiotics, antiviral (except antiviral therapy directed at hepatitis B) or antifungal agents. Such infection must be fully resolved prior to randomization.
* Ascites requiring paracentesis within 14 days prior to randomization.
* Uncontrolled hypertension, defined as an average systolic blood pressure > 159 mmHg or diastolic > 99 mmHg despite optimal treatment (measured according European Society of Hypertension/European Society of Cardiology [ESH / ESC] 2013 guidelines[65].
* History of stroke or intracranial hemorrhage within 6 months prior to randomization.
* Known interstitial lung disease.
* Infiltrative pulmonary disease, known pulmonary hypertension.
* Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal.
* Known severe persistent asthma within the past 2 years (see also https://www.nhlbi.nih.gov/files/docs/guidelines/asthsumm.pdf), or currently has uncontrolled asthma of any classification or at time of screening has an FEV1 of < 50% of predicted normal.
* Autologous or allogeneic stem cell transplant less than 100 days prior to randomization.
* Vaccination with live attenuated vaccines within 30 days prior to randomization.
* Patients who require strong or moderate inducers or inhibitors for cytochrome P450, family 3 or subfamily A (CYP3A).
* Patients who have an uncontrolled bleeding disorder or require an anticoagulant (e.g. warfarin or other vitamin K antagonists; novel oral anticoagulants (NOACs) are allowed) at time of screening.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or sponsor, if consulted, would pose a risk to patient safely or interfere with the study evaluation, procedures or completion.
* Patient is a woman who is pregnant or breastfeeding (and do not consent to discontinue breast-feeding) or planning to become pregnant while enrolled in this study or within 6 months after the last study treatment.
* Vulnerable patients, e.g. patients who are incapable of giving informed consent (severe dementia or psychosis, patients kept in detention).
* Participation in another interventional clinical study within 30 days before randomization in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
CR/VGPR | 12 months
  Primary endpoint is the rate of CR or VGPR 12 months after the start of treatment using the response criteria updated at the Sixth IWWM (CR/VGPR).

SECONDARY OUTCOMES:
Response rate | 12/ 24 months
  The response rates (CR, VGPR, PR, MR) and overall response rate (CR, VGPR, PR, MR) are evaluated 12 and 24 months after the start of treatment.
Best response | 12 months
  Best response (at least achieving a MR) is determined in the time interval from the start of induction therapy to end of follow-up.
Time to best response | 12 months
  Time to best response is defined as the time from the start of induction to best response the patient achieves (CR, VGPR, PR, MR).
Time to first response | 12 months
  Time to first response is defined as the time from the start of induction to first response (MR, PR, VGPR or CR).
Time to treatment failure (TTF) | 7 years
  TTF is defined as the time of start of induction treatment to discontinuation of therapy for any reason including death from any cause, progression, toxicity or add-on of new anti-cancer therapy. Patients alive without progression and relapse will be censored at the latest tumor assessment date.
Remission duration (RD) | 7 years
  Remission duration will be calculated in patients with response (CR, VGPR, PR, MR) from the date of response to the date of progression, relapse or death from any cause. Patients alive without progression and relapse will be censored at the latest tumor assessment date.
Progression Free Survival (PFS) | 7 years
  PFS will be calculated from the date of start of treatment to the following events: the date of progression (as defined in Appendix A) and the date of death if it occurred earlier. Patients alive without progression and relapse will be censored at the latest tumor assessment date.
Cause specific survival (CSS) | 7 years
  Cause specific survival is defined as the period from the start of induction treatment to death from lymphoma or lymphoma related cause; death unrelated to WM is considered as a competing event.
Overall survival (OS) | 7 years
  Overall survival is defined as the period from the start of induction treatment to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.
Rate of Adverse Events (safety) | 7 years
  Number of adverse events and comparison of adverse event rate in both treatment arms.
Changes in Quality of Life | 7 years
  Changes in quality of life will be assessed by the FACT-Lym questionnaire and compared in both treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Buske, MD, Study Chair — University of Ulm
Locations (20):
- Austria (2):
  - Uniklinikum Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Germany (17):
  - Vivantes Klinikum am Urban, Berlin
  - Ev. Diakoniekrankenhaus, Bremen
  - Kath. St.-Johannes-Gesellschaft Dortmund gGmbH, Dortmund
  - Gemeinschaftspraxis Mohm / Prange-Krex, Dresden
  - OncoResearch Lerchenfeld GmbH, Hamburg
  - MediProject Onkologisches Ambulanzzentrum Hannover, Hanover
  - Praxis für Hämatologie und Onkologie, onkologische Tagesklinik-VK&K Studien GbR, Landshut
  - Praxis Dr. Vehling-Kaiser, Landshut
  - Rotkreuzklinikum München, Munich
  - Hämatologie/Onkologie München Pasing MVZ GmbH, Munich
  - Kliniken Ostalb, Staufenklinikum Schw. Gmuend, Mutlangen
  - Friedrich-Ebert-Krankenhaus, Neumünster
  - Bruederkrankenhaus St. Josef, Paderborn
  - Universitätsmedizin Rostock, Rostock
  - Klinikum Mutterhaus Mitte Trier gGmbh Studienzentrum, Trier
  - University Hospital Ulm, Ulm
  - Hämatologisch-Onkologische Schwerpunktpraxis Drs. Schöttker & Pretscher, Würzburg
- Alexandra Hospital, Athens, Greece